CLINICAL TRIAL: NCT00403013
Title: Axillary Plexus Block for Perioperative Analgesia in Patients Scheduled for Elective Surgery of the Shoulder: Influence of Lateral, Head-Down Position
Brief Title: Plexus Anesthesia in Lateral, Head-Down Position for Elective Surgery of the Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principle Investigator, Department of Anesthesiology and Intensive Care, University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-AnIt-06
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Shoulder Surgery
Keywords: nerve block/*methods; Anesthetics, Local/pharmacokinetics; *Brachial Plexus
MeSH Terms: interventions — Patient Positioning; Anesthesia

ARMS (2):
- 1 (Experimental): lateral, head-down position during axillary plexus block
  Interventions: Procedure: Positioning and anesthesia
- 2 (Active Comparator): standard position during axillary plexus block
  Interventions: Procedure: Positioning and anesthesia

INTERVENTIONS:
Procedure: Positioning and anesthesia — Positioning during axillary plexus block

SUMMARY:
The purpose of this study is to determine whether the axillary plexus block performed in lateral, head down position is effective in the perioperative analgesia in patients scheduled for elective surgery of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective surgery of the shoulder

Exclusion Criteria:

* lateral, head down position not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) score | 8 hours after start of axillary plexus block
VAS Score | 24 hours after start of axillary plexus block

SECONDARY OUTCOMES:
Opioid consumption | intraoperatively
Patient comfort | six months after surgery
Opioid consumption | during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: T Weber, MD, Principal Investigator — Department of Anesthesiology and Intensive Care, University Hospital Muenster
Locations (1):
- Department of Anesthesiology and Intensive Care, University Hospital Muenster, Münster, Germany

REFERENCES:
- [Background] Orlowski O, Bullmann V, Vieth V, Filler T, Osada N, Van Aken H, Weber TP. Perivascular axillary brachial plexus block and patient positioning: the influence of a lateral, head-down position. Anaesthesia. 2006 Jun;61(6):528-34. doi: 10.1111/j.1365-2044.2006.04618.x. PMID 16704585